CLINICAL TRIAL: NCT04383639
Title: Evaluation of Postprandial Effects of High Molecular Weight Polyphenols in Subjects With Type 2 Diabetes
Brief Title: Cocoa/Carob Polyphenols and Postprandial Changes in Type 2 Diabetes
Acronym: CACAOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Jara Pérez-Jiménez, Principal Investigator, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RTI2018DIABE
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
Keywords: Polyphenols; Type 2 diabetes; Cocoa; Carob; Postprandial response; Insulin resistance; Microbial metabolites
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Breakfast; locust bean gum

STUDY DESIGN:
Intervention Model Description: A: control period; B: mixture of cocoa and carob consumed together with breakfast; C: mixture of cocoa and carob consumed 10 h before breakfast. All the subjects will pass the three treatments, in randomized order. The three periods will be separated by a two weeks washing period.
Who Masked: Outcomes Assessor
Masking Description: Since no placebo was found, the subjects will know the treatment they are receiving in each case. Nevertheless, the outcome assessor will not know to which treatment corresponds each sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator): All subjects will receive a high-fat high-sugar breakfast in three different days. They will not consume any additional product (1), they will receive the mixture of coca and carob together with breakfast (2) or they will receive the mixture of coca and carob 10 h before breakfast (3).
  Interventions: Other: No product (A)/mixture of coca and carob together with breakfast (B)/mixture of coca and carob 10 h before breakfast (C)
- 2 (Experimental): All subjects will receive a high-fat high-sugar breakfast in three different days. They will not consume any additional product (1), they will receive the mixture of coca and carob together with breakfast (2) or they will receive the mixture of coca and carob 10 h before breakfast (3).
  Interventions: Other: No product (A)/mixture of coca and carob together with breakfast (B)/mixture of coca and carob 10 h before breakfast (C)
- 3 (Experimental): All subjects will receive a high-fat high-sugar breakfast in three different days. They will not consume any additional product (1), they will receive the mixture of coca and carob together with breakfast (2) or they will receive the mixture of coca and carob 10 h before breakfast (3).
  Interventions: Other: No product (A)/mixture of coca and carob together with breakfast (B)/mixture of coca and carob 10 h before breakfast (C)

INTERVENTIONS:
Other: No product (A)/mixture of coca and carob together with breakfast (B)/mixture of coca and carob 10 h before breakfast (C) — The subjects will receive, after overnight fasting, a high-fat high-sugar breakfast. In treatment A, they will not receive any additional product; in treatment B, they will receive at the same time a mixture of coca and carob; in treatment C, they will receive the mixture of coca and carob 10 h before breakfast. A total of 6 blood samples will be collected during each visit: 0-30-60-120-180-240-270 min. Urine samples will be collected during the permanence of the subjects in the Unit of Human Nutrition. Feces will be collected the first time they are generated after treatments A and C. Both interventions will be separated by two weeks. Subjects will be instructed not to modify their dietary habits during the development of the study, but during the 72 h before each visit they will have to restrict the intake of polyphenol-rich foods (a detailed list will be provided).

SUMMARY:
The aim of this is study is to evaluate the effects of a single intake of a mixture of cacao and carob (rich in high molecular weight polyphenols) in postprandial metabolism in subjects with type 2 diabetes. Studies on the effects of polyphenols on postprandial (glucidic and lipidic) metabolism have commonly been performed in animal models and have used food extracts, ignoring high molecular weight polyphenols as relevant bioactive compounds. In this study, the potential of this kind of polyphenols for regulating postprandial disturbances in type 2 diabetes subjects, since these alterations increased the cardiovascular risk in these subjects, will be evaluated. The study has been designed in order to differentially evaluate the effect of intact polyphenols and that of microbial-derived phenolic metabolites.

DETAILED DESCRIPTION:
Twenty-five subjects with a recent diagnosis of type 2 diabetes will be recruited. Detailed inclusion and exclusion criteria are provided below.

The whole intervention has been divided in 3 treatments A, B and C, performed every 2 weeks in randomized order for each subject. In every treatment, subjects will attend to the Unit of Human Nutrition of the ICTAN-CSIC in fasting state and they will receive a high-sugar high-fat breakfast. Treatment A will be used as control and will only consist of breakfast. Treatment B is characterized by the administration of a mixture of cocoa and carob solved in milk together with breakfast. In treatment C, volunteers will consume the same amount of product 10 hours before attending to their visit, where the breakfast will be administrated once again. Food and drinks provided in the three visits (including milk used in treatment B) will be similar. The aim of treatment B is to elucidate the role of intact polyphenols, while treatment C will evaluate the effect of microbial-derived polyphenol metabolites.

Blood samples will be collected before breakfast and at times 60-120-180-240-270 min. Urine will be collected during their permanence at the Unit of Human nutrition of the ICTAN-CSIC. Feces will be collected as soon as they are generated after receiving treatments A and C. The following determinations will be performed in blood samples collected at different periods: glucose, insulin, triglycerides, uric acid, GLP-1, hepatic enzymes. Urine and feces will be used to evaluate phenolic metabolites. Additionally, a satiety test will be provided. It is expected that cocoa and carob supplementation, as compared to the control treatment, causes significant modifications in all the parameters indicated. Nevertheless, the primary outcome of this study is the decrease in postprandial insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes during the last 2 years and current treatment with metformin
* Overweight or obesity (IMC = 26-40 kg/m2)

Exclusion Criteria:

* Subjects with a pharmaceutical treatment set to modify blood pressure, lipid profile or glucose.
* Subjects with diagnoses of cardiovascular diseases or thyroid diseases.
* Values above the following ones: glucose, > 125 mg/dL; triglycerides, > 350 mg/dL; total cholesterol, > 280 mg/dL; systolic blood pressure, > 150 mmHg; diastolic blood pressure, > 100 mmHg
* Previous bariatric surgery.
* Volunteers currently participating in other studies or weight loss plans.
* Pregnant or breastfeeding women.
* Adherence to vegetarian diets or usual consumption of dietary supplements.
* Intolerance or allergy to some of the foods provided in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Postprandial insulin | Up to two months
  Changes of postprandial insulin as result of supplementation with cocoa and carob

SECONDARY OUTCOMES:
Postprandial glucose | Up to four months
  Changes of blood glucose as result of supplementation with cocoa and carob.
Postprandial triglycerides | Up to four months
  Changes of blood triglycerides as result of supplementation with cocoa and carob.
Postprandial uric acid | Up to four months
  Changes of blood uric acid as result of supplementation with cocoa and carob.
Postprandial GLP-1 | Up to five months
  Changes of blood GLP-1 as result of supplementation with cocoa and carob.
Postprandial phenolic metabolites | Up to six months
  Changes of urinary and fecal phenolic metabolites as result of supplementation with cocoa and carob.
Satiety measured by a Visual Analogue Scale (see "Description" for details) | Up to three months
  Changes of satiety as result of supplementation with cocoa and carob. This will be determined by the CSS, composite satiety score. This is a value obtained from a formula once the subject has filled in, in a visual analogue scale, the answer to different questions regarding hunger and satiety. The answers go from 1 to 10 (each mark corresponding to a similar distance in the scale). The final CSS value goes also from 1 to 10, with 1 meaning the lowest satiety and 10 meaning the highest one.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food Science, Technology and Nutrition, National Research Council (ICTAN-CSIC), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided